CLINICAL TRIAL: NCT03067311
Title: Targeting Stress Reactivity in Schizophrenia: Integrated Coping Awareness Therapy (I-CAT)
Brief Title: Targeting Stress Reactivity in Schizophrenia: Integrated Coping Awareness Therapy
Acronym: I-CAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-1173; 4R33MH100250-03 (NIH)
Record Dates: First submitted 2017-02-16; First posted 2017-03-01 (Actual); Results first posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2020-05

CONDITIONS: Schizophreniform Disorders
MeSH Terms: conditions — Psychotic Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-CAT (Experimental): A novel therapeutic intervention combining strategies to improve stress reactivity and increase meaningful coping given by trained clinicians.
  Interventions: Behavioral: I-CAT
- Treatment as Usual (Active Comparator): Usual treatment provided at the University of North Carolina at Chapel Hill (UNC) Outreach and Support Intervention Services (OASIS) Clinic by trained clinicians.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: I-CAT — I-CAT is a novel therapeutic intervention combining mindfulness and meditation strategies to improve stress reactivity and increase meaningful coping, as well as a range of possible proximal (e.g. autonomic, endocrine, immune indices of stress reactivity, symptom severity) and distal measures (function, relapse, quality of life).
  Arms: I-CAT
Behavioral: Treatment as Usual — Treatment as usual defined by participant clinician at OASIS clinic.
  Arms: Treatment as Usual

SUMMARY:
To test the feasibility of a clinical trial implementing I-CAT, a novel therapeutic intervention combining strategies to improve stress reactivity and increase meaningful coping, as well as a range of possible proximal (e.g. autonomic, endocrine, immune indices of stress reactivity, symptom severity) and distal measures (function, relapse, quality of life) for 40 people with first episode psychosis in the context of a small randomized controlled trial.

DETAILED DESCRIPTION:
Schizophrenia is one of the most devastating disorders that often results in a lack of functional recovery. Current treatments focused on remediating symptoms have shown only small successes in a return to functioning despite evidence of a dysregulated stress response. There is a fundamental gap in understanding the impact of allostatic overload in persons with schizophrenia that the investigators theorize is associated with deficits in functioning and with an increased vulnerability and relapse risk. The long-term goal is to test an intervention aimed at improving stress reactivity. The objective in this application is to develop and test the feasibility of a novel therapeutic intervention combining strategies to improve stress reactivity and increase meaningful coping. The central hypothesis is that an intervention that improves stress reactivity as measured proximally by endocrine, immune, and autonomic indices will result in improved adaptive capacity, better role functioning, reduced risk of relapse, and decreased likelihood of disability for people in the early stages of schizophrenia.

The rationale for the proposed research is that stress reactivity may be a modifiable risk factor underlying functional deficits in schizophrenia. The intervention integrates two treatment approaches. The first is based on research showing that mindfulness meditation practice is associated with alterations in the neural processing of stressful events and targets adaptive responses to stress. The second focuses on providing a buffer against stress by using the self-generation of adaptive emotions with a positive psychology intervention, which is potentially associated with building protective social resources. These complimentary interventions provide a comprehensive synergistic approach for this population that could lead to more adaptive coping responses and create a buffer against stress

ELIGIBILITY:
Inclusion Criteria:

* meets Diagnostic and Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for schizophrenia spectrum disorder according diagnostic checklist completed by individual's clinician
* age 15 to 35, both genders, and any ancestry
* currently receiving services from UNC OASIS, Schizophrenia Treatment and Evaluation Program (STEP), or a community clinic
* willing and able to provide informed consent

Exclusion Criteria:

* greater than 8 years of antipsychotic and/or psychological treatment for psychosis
* Intelligence Quotient (IQ) less than 80
* low stress level as reported by clinician or participant
* meets criteria for current substance dependence
* been hospitalized in the past month
* actively practicing meditation in the past year

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David L Penn, PhD, Principal Investigator — The Unviersity of North Carolina at Chapel Hill; Diana Perkins, MD, Principal Investigator — The Unviersity of North Carolina at Chapel Hill; Piper S Meyer-Kalos, PhD, Principal Investigator — Minnesota Center for Chemical and Mental Health
Locations (4):
- United States (4):
  - UNC OASIS Carrboro, Carrboro, North Carolina
  - UNC STEP, Carrboro, North Carolina
  - UNC Oasis Wake, Raleigh, North Carolina
  - UNC Wake STEP, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment as Usual: Usual treatment provided at the University of North Carolina at Chapel Hill (UNC) OASIS Clinics by trained clinicians.
  Treatment as Usual: Treatment as usual defined by participant clinician at OASIS clinic.
Period: Overall Study
Arm/Group | I-CAT | Treatment as Usual
Started | 19 | 19
Completed | 17 | 17
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Moved away | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment as Usual: Usual treatment provided at the UNC OASIS Clinics by trained clinicians.
  Treatment as Usual: Treatment as usual defined by participant clinician at OASIS clinic.
- Total: Total of all reporting groups
Arm/Group | I-CAT | Treatment as Usual | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 19 | 38
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.6 (4.3) | 24.9 (3.9) | 24.3 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 15 | 18 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 11 | 14 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 19 | 38
WASI-II Intelligence Quotient (IQ) Score [Mean (Standard Deviation); unit: t-score] — Wechsler Abbreviated Scale of Intelligence - 2nd Edition (WASI-II) is a standardized test of intelligence consisting of Matrix Reasoning, Vocabulary, Similarities, and the Block Design subtests with a total score that is converted to a standard t-score (possible range 40 - 160). A t-score of 50 is equal to the mean of the population with a standard deviation of 10. Scores less than 50 reflect scores less than the mean of the population whereas scores greater than 50 reflect scores more than the mean of the population. Higher scores indicate higher levels of intelligence.
  t-score | 107.7 (14.1) | 111.5 (12) | 109.6 (13.05)
Duration of Illness [Mean (Standard Deviation); unit: years] — Duration of Illness is defined as the years between study enrollment and initial schizophrenia spectrum disorder (SSD) diagnosis (range 0 - 9 for the current study).
  years | 1.7 (1.5) | 1.8 (2) | 1.8 (1.8)
PANSS Total [Mean (Standard Deviation); unit: units on a scale] — The Positive and Negative Syndrome Scale (PANSS) assessed current symptoms. PANSS items are rated on a seven-point scale with higher scores reflecting more severe symptoms (ICCs for study assessors >.90). Items are summed for a total score (range 30 - 210).
  units on a scale | 62.3 (17.2) | 58.4 (16) | 60.4 (16.6)
mDES - Positive Emotions [Mean (Standard Deviation); unit: units on a scale] — The modified self-report Differential Emotion Scale (mDES) assessed the frequency of experiencing discrete emotions from the previous week. Items are endorsed on a five-point scale indicating frequency (0 = not at all, 4 = most of the time). Items are summed to yield positive (mDES - Positive) and negative emotion (mDES - Negative) subscales (range for both 0-40). Higher scores on the positive subscale indicate more positive emotions.
  units on a scale | 21.3 (6.9) | 20.9 (9.3) | 21.1 (8.1)
mDES - Negative Emotions [Mean (Standard Deviation); unit: units on a scale] — The modified self-report Differential Emotion Scale (mDES) assessed the frequency of experiencing discrete emotions from the previous week. Items are endorsed on a five-point scale indicating frequency (0 = not at all, 4 = most of the time). Items are summed to yield positive (mDES - Positive) and negative emotion (mDES - Negative) subscales (range for both 0-40). Higher scores on the negative subscale indicate more negative emotions.
  units on a scale | 15.6 (8.7) | 18.2 (10.6) | 16.9 (9.65)
Quality of Life Scale [Mean (Standard Deviation); unit: units on a scale] — The Quality of Life Scale (QLS) is a semi-structured 7-item interview with sub scales, including active acquaintances, social initiatives, occupational role functioning, degree of motivation, anhedonia, commonplace objects, and capacity for empathy. The 7-items are rated on a 7-point scale with higher ratings reflecting less impaired functioning (total range 7-49).
  units on a scale | 26 (8.3) | 25.3 (7.2) | 25.7 (7.8)
First Episode Social Functioning Scale [Mean (Standard Deviation); unit: units on a scale] — The First Episode Social Functioning Scale (FESFS) is a 42-item self-report measure assessing social functioning in early SSD. The FESFS includes a total score and eight subscales assessing: independent living skills, interacting with people in different contexts, social activities, intimacy, friendships, family relations, work, and school. Domain scores are averaged with higher scores reflecting better perceived functioning (range 0-4).
  units on a scale | 3 (0.4) | 3.2 (0.5) | 3.1 (0.45)
Perceived Stress Scale [Mean (Standard Deviation); unit: units on a scale] — The Perceived Stress Scale (PSS) is a ten-item self-report measure of the degree to which daily situations from the past week are perceived as stressful, unpredictable, uncontrollable, as well as how "overloaded" individuals feel (0 = never, 4 = very often). Items are summed for a total score (range 0 - 40) with higher scores indicating more perceived stress.
  units on a scale | 18.8 (6.3) | 20.9 (8.5) | 19.9 (7.4)
Daily Stress Inventory [Mean (Standard Deviation); unit: units on a scale] — The Daily Stress Inventory (DSI) is a 58-item self-report measure assessing the frequency and intensity of stressful events within the past 24-hours. If an event is endorsed, participants rate the amount of stress the event caused (0 = did not occur, 1 = occurred but was not stressful to 7 = occurred and caused me to panic). The DSI yields an average impact rating (AIR; average impact of ratings given items endorsed [sum/frequency]; range 1-7) with higher scores reflecting higher levels of stress experienced.
  units on a scale | 3.0 (1.3) | 2.9 (1.2) | 2.95 (1.25)
Five Facets of Mindfulness Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The Five Facet Mindfulness Questionnaire (FFMQ) is a 39-item self-report measure assessing facets of being mindful in daily life (i.e., observing, describing, acting with awareness, non-reactivity to inner experience, and non-judging of inner experience). Items are endorsed on a five-point scale (1 = never or rarely true to 5 = very often or always true) and averaged for a total score (range 1-5) with higher scores reflecting greater mindfulness abilities.
  units on a scale | 3 (0.4) | 3 (0.6) | 3 (0.5)
Self-Compassion Scale [Mean (Standard Deviation); unit: units on a scale] — The Self-Compassion Scale Short Form (SCS) is a 12-item self-report measure of self-compassion. SCS items are endorsed on a five-point scale (1 = almost never to 5 = almost always) and are summed for a total score (range 12 - 60) with higher scores indicating higher levels of self-compassion.
  units on a scale | 34.7 (7) | 35.7 (9.7) | 35.2 (8.35)
Perceived Well-Being Scale [Mean (Standard Deviation); unit: units on a scale] — The Psychological Well-Being Scale (PWB) is a 54-item self-report measure with items endorsed on a seven-point scale (1 = strongly disagree to 6 = strongly agree). Items are summed for a total score (range 54 - 324) with higher scores indicating better psychological well-being.
  units on a scale | 207.9 (36.8) | 209.32 (46.8) | 208.61 (41.8)

OUTCOME MEASURES:

1. Primary Outcome: Change Over Time on the mDES - Positive
Description: The modified self-report Differential Emotion Scale (mDES) assessed the frequency of experiencing discrete emotions from the previous week. Items are endorsed on a five-point scale indicating frequency (0 = not at all, 4 = most of the time). Items are summed to yield positive (mDES - Positive) and negative emotion (mDES - Negative) subscales (range for both 0-40). Higher scores on the positive subscale indicate more positive emotions. Assessed at 4.5 months, 9 months, 12 months.
Time Frame: Baseline, 4.5, 9, and 12 months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | I-CAT | Treatment as Usual
Number analyzed (Participants) | 17 | 17
units on a scale
  4.5 months change from baseline | 0.35 (0.19) | 0.42 (0.20)
  9 months change from baseline | 0.62 (0.19) | 0.25 (0.19)
  12 months change from baseline | 0.28 (0.19) | 0.38 (0.21)

2. Primary Outcome: Change Over Time on the mDES - Negative
Description: The modified self-report Differential Emotion Scale (mDES) assessed the frequency of experiencing discrete emotions from the previous week. Items are endorsed on a five-point scale indicating frequency (0 = not at all, 4 = most of the time). Items are summed to yield positive (mDES - Positive) and negative emotion (mDES - Negative) subscales (range for both 0-40). Higher scores on the negative subscale indicate more negative emotions. Assessed at 4.5 months, 9 months, 12 months.
Time Frame: Baseline, 4.5, 9, and 12 months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | I-CAT | Treatment as Usual
Number analyzed (Participants) | 17 | 17
units on a scale
  4.5 months change from baseline | 0.01 (0.17) | -0.38 (0.20)
  9 months change from baseline | -0.27 (0.17) | -0.19 (0.19)
  12 months change from baseline | -0.01 (0.19) | -0.24 (0.20)

3. Primary Outcome: Change Over Time on the QLS
Description: The Quality of Life Scale (QLS) is a semi-structured 7-item interview with sub scales, including active acquaintances, social initiatives, occupational role functioning, degree of motivation, anhedonia, commonplace objects, and capacity for empathy. The 7-items are rated on a 7-point scale with higher ratings reflecting less impaired functioning (total range 7-49). Assessed at 4.5 months, 9 months, 12 months.
Time Frame: Baseline, 4.5, 9, and 12 months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | I-CAT | Treatment as Usual
Number analyzed (Participants) | 17 | 17
units on a scale
  4.5 months change from baseline | 0.10 (0.16) | 0.36 (0.78)
  9 months change from baseline | 0.26 (0.16) | 0.28 (0.18)
  12 months change from baseline | 0.74 (0.16) | 0.91 (0.18)

4. Primary Outcome: Change Over Time on the FESFS
Description: The First Episode Social Functioning Scale (FESFS) is a 42-item self-report measure assessing social functioning in early SSD. The FESFS includes a total score and eight subscales assessing: independent living skills, interacting with people in different contexts, social activities, intimacy, friendships, family relations, work, and school. Domain scores are averaged with higher scores reflecting better perceived functioning (range 0-4). Assessed at 4.5 months, 9 months, 12 months.
Time Frame: Baseline, 4.5, 9, and 12 months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | I-CAT | Treatment as Usual
Number analyzed (Participants) | 17 | 17
units on a scale
  4.5 months change from baseline | -0.07 (0.14) | 0.04 (0.16)
  9 months change from baseline | 0.22 (0.15) | 0.20 (0.15)
  12 months change from baseline | 0.40 (0.15) | 0.33 (0.17)

5. Primary Outcome: Change Over Time on the PSS
Description: The Perceived Stress Scale (PSS) is a ten-item self-report measure of the degree to which daily situations from the past week are perceived as stressful, unpredictable, uncontrollable, as well as how "overloaded" individuals feel (0 = never, 4 = very often). Items are summed for a total score (range 0 - 40) with higher scores indicating more perceived stress. Assessed at 4.5 months, 9 months, 12 months.
Time Frame: Baseline, 4.5, 9, and 12 months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | I-CAT | Treatment as Usual
Number analyzed (Participants) | 17 | 17
units on a scale
  4.5 months change from baseline | -0.26 (0.19) | -0.46 (0.23)
  9 months change from baseline | -0.36 (0.19) | -0.44 (0.20)
  12 months change from baseline | -0.16 (0.20) | -0.52 (0.22)

6. Primary Outcome: Change Over Time on the DSI
Description: The Daily Stress Inventory (DSI) is a 58-item self-report measure assessing the frequency and intensity of stressful events within the past 24-hours. If an event is endorsed, participants rate the amount of stress the event caused (0 = did not occur, 1 = occurred but was not stressful to 7 = occurred and caused me to panic). The DSI yields an average impact rating (AIR; average impact of ratings given items endorsed [sum/frequency]; range 1-7) with higher scores indicating more daily stress. Assessed at 4.5 months, 9 months, 12 months.
Time Frame: Baseline, 4.5, 9, and 12 months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | I-CAT | Treatment as Usual
Number analyzed (Participants) | 17 | 17
units on a scale
  4.5 months change from baseline | 0.09 (0.23) | -0.09 (0.23)
  9 months change from baseline | 0.46 (0.22) | -0.12 (0.23)
  12 months change from baseline | -0.41 (0.24) | -0.51 (0.25)

7. Primary Outcome: Change Over Time on Salivary Cortisol Levels
Description: Salivary cortisol levels were collected as a measure of psychological stress.
Time Frame: Baseline, 9 months
Population: Saliva samples unable to be collected from all participants.
Measure: Least Squares Mean (Standard Error); unit: ug/dL
Arm/Group | I-CAT | Treatment as Usual
Number analyzed (Participants) | 17 | 12
ug/dL | 0.0254 (0.0240) | -0.0124 (0.0274)

8. Secondary Outcome: Change Over Time on the PANSS Total Score
Description: The Positive and Negative Syndrome Scale (PANSS) assessed current symptoms. PANSS items are rated on a seven-point scale with higher scores reflecting more severe symptoms (ICCs for study assessors >.90). Items are summed for a total score (range 30 - 210). Assessed at 4.5 months, 9 months, 12 months.
Time Frame: Baseline, 4.5, 9, and 12 months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | I-CAT | Treatment as Usual
Number analyzed (Participants) | 17 | 17
units on a scale
  4.5 months change from baseline | -0.49 (0.15) | -0.29 (0.16)
  9 months change from baseline | -0.81 (0.15) | -0.29 (0.16)
  12 months change from baseline | -1.00 (0.15) | -0.66 (0.17)

9. Secondary Outcome: Change Over Time on the FFMQ
Description: The Five Facet Mindfulness Questionnaire (FFMQ) is a 39-item self-report measure assessing facets of being mindful in daily life (i.e., observing, describing, acting with awareness, non-reactivity to inner experience, and non-judging of inner experience). Items are endorsed on a five-point scale (1 = never or rarely true to 5 = very often or always true) and averaged for a total score (range 1-5) with higher scores indicating greater mindfulness ability. Assessed at 4.5 months, 9 months, 12 months.
Time Frame: Baseline, 4.5, 9, and 12 months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | I-CAT | Treatment as Usual
Number analyzed (Participants) | 17 | 17
units on a scale
  4.5 months change from baseline | 0.18 (0.144) | 0.51 (0.15)
  9 months change from baseline | 0.35 (0.14) | 0.26 (0.14)
  12 months change from baseline | 0.26 (0.14) | 0.13 (0.15)

10. Secondary Outcome: Change Over Time on the SCS
Description: The Self-Compassion Scale Short Form (SCS) is a 12-item self-report measure of self-compassion. SCS items are endorsed on a five-point scale (1 = almost never to 5 = almost always) and are summed for a total score (range 12 - 60) with higher scores indicating higher levels of self-compassion. Assessed at 4.5 months, 9 months, 12 months.
Time Frame: Baseline, 4.5, 9, and 12 months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | I-CAT | Treatment as Usual
Number analyzed (Participants) | 17 | 17
units on a scale
  4.5 months change from baseline | -0.06 (0.18) | 0.30 (0.20)
  9 months change from baseline | 0.11 (0.18) | 0.27 (0.19)
  12 months change from baseline | 0.04 (0.19) | 0.13 (0.20)

11. Secondary Outcome: Change Over Time on the PWB
Description: The Psychological Well-Being Scale (PWB) is a 54-item self-report measure with items endorsed on a seven-point scale (1 = strongly disagree to 6 = strongly agree). Items are summed for a total score (range 54 - 324) with higher scores indicating better psychological well-being. Assessed at 4.5 months, 9 months, 12 months.
Time Frame: Baseline, 4.5, 9, and 12 months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | I-CAT | Treatment as Usual
Number analyzed (Participants) | 17 | 17
units on a scale
  4.5 months change from baseline | 0.21 (0.14) | 0.17 (0.15)
  9 months change from baseline | 0.36 (0.14) | -0.01 (0.15)
  12 months change from baseline | 0.29 (0.14) | 0.12 (0.16)

12. Secondary Outcome: Respiratory Sinus Arrhythmia
Description: Index of heart rate variability assessed as the ratio of low-to-high frequencies in the respiratory-cardiac power spectrum. Mean level respiratory sinus arrhythmia (RSA) derived from heart rate monitor worn while participants engaged in a 5-minute mindfulness exercise.
Time Frame: 9 months
Population: Data not available for all participants due to device technical issues or post-treatment appointment completed remotely.
Measure: Least Squares Mean (Standard Error); unit: ln(msec)^2
Arm/Group | I-CAT | Treatment as Usual
Number analyzed (Participants) | 9 | 11
ln(msec)^2 | 4.58 (0.520) | 6.15 (0.562)

ADVERSE EVENTS:
Time Frame: From baseline to study follow-up, a total of approximately 12 months.
Arm/Group | I-CAT | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 3/19 | 2/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | I-CAT (N=19) | Treatment as Usual (N=19)
Increased psychiatric symptoms (General disorders) | 1 (1) | 2 (4) — Hospitalization due to increased psychiatric symptoms.
Discontinued medication (General disorders) | 1 (1) | 0 (0) — Participant discontinued psychiatric medication precipitating an increase in psychiatric symptoms, specifically suicidal ideation, which necessitated hospitalization
Dyskinesia (General disorders) | 1 (1) | 0 (0) — Participant experienced dyskinesia precipitating hospitalization

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/11/NCT03067311/Prot_SAP_000.pdf